CLINICAL TRIAL: NCT06843161
Title: Retraining Automatic Attitudes Towards Physical Activity and Sedentary Behaviour in Adults 60 Years of Age or Older
Brief Title: Robot-based Intervention to Improve Physical Activity in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Banting Research Foundation (Unknown); Mitacs (Industry); Perley Health (Unknown)
Responsible Party: Principal Investigator, Kayne Park, Principal Investigator, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-01-25-11168
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Physical Inactivity; Aging; Sedentary Behaviors; Bias, Implicit; Cognition
MeSH Terms: conditions — Sedentary Behavior; Bias, Implicit

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group: Responses Biased towards Visual Stimulus (Experimental): Successfully recruited individuals will be performing the JOGGNG Task on the Kinarm Endpoint Laboratory. This task requires participants to quickly make a reaching movement to manipulate a virtual avatar that is jogging across a field. During this, a frisbee will move towards the avatar and will tilt clockwise or counterclockwise. Participants have been instructed to either reach quickly to grab the frisbee from the air during clockwise tilts or to not move during counterclockwise tilts. This tilt/movement associated is reversed to control for potential bias in tilt angle and movement. An image of physical activity or sedentary behaviour will appear inside of the frisbee but participants are not told that it is associated with any of the tilts. For the Interventional Group, the tilt associated with movement will have an image of physical activity appear 90% of the time and the tilt associated with no movement will have an image of sedentary behaviour 90% of the time.
  Interventions: Device: The jog or ground go no go task for retraining automatic bias
- Control Group: Responses Randomly Assigned to Visual Stimulus (Sham Comparator): Recruited participants will be performing the JOGGNG Task on the Kinarm Endpoint Laboratory. This task requires participants to quickly make a reaching movement to manipulate a virtual avatar that is jogging across a field. During this, a frisbee will move towards the avatar and will tilt clockwise or counterclockwise. Participants have been instructed to either reach quickly to grab the frisbee from the air during clockwise tilts or to not move during counterclockwise tilts. This tilt/movement associated is reversed to control for potential bias in tilt angle and movement. An image of physical activity or sedentary behaviour will appear inside of the frisbee but participants are not told that it is associated with any of the tilts. For the Control Group, the tilt associated with movement will have an image of physical activity appear 50% of the time and the tilt associated with no movement will have an image of sedentary behaviour 50% of the time.
  Interventions: Device: The jog or ground go no go task for retraining automatic bias

INTERVENTIONS:
Device: The jog or ground go no go task for retraining automatic bias — Recruited participants will be performing the JOGGNG Task on the Kinarm Endpoint Laboratory. This task requires participants to control a robotic handle to manipulate a virtual avatar that looks as if it is jogging across a field. During the jogging, a frisbee will appear and quickly move towards the avatar, eventually tilting clockwise or counterclockwise. Participants are required to either reach quickly to grab the frisbee from the air during clockwise tilts or to not move during counterclockwise tilts. This tilt/movement associated is reversed to control for a potential bias in tilt angle and movement. An image of physical activity or sedentary behaviour will appear inside of the frisbee but participants are not told that it is associated with any of the tilts. Each trial consists of one frisbee and participants will complete a total of 3 blocks of 360 trials each which will take approximately 30 minutes to complete.

SUMMARY:
Physical inactivity is considered a global pandemic negatively impacting the health of over 60% of older adults in America. Interventions aimed at improving physical activity in older adults focus on training reflective processes such as providing information on health benefits of physical activity. These interventions generally find that participants improved their intentions to be physically active rather than supporting actual change in behaviours to become physically active.

There is growing support for the idea that human behaviour is the result of a combination of quick automatic processes and slower reflective processes. Interventional studies have used cognitive bias modification tasks that target the quick automatic processes to retrain participant's bias. Such studies find that participant's bias towards diet, alcohol, and phobias can be altered using these cognitive bias modification tasks.

In this study, the investigators developed a new training task using a robotic device that aims to retrain automatic bias towards physical activity and sedentary behaviours. The robotic device allows greater immersive environments for participants to interact with and be more engaged with the cognitive bias modification task. This interventional study is testing whether this new robot-based training and the protocol for assessing physical activity is feasible for retraining older adults' bias towards physical activity and sedentary behaviour. Participants will be examined on their daily physical activity using an accelerometer, their physical ability using functional tests, and their perceptions on physical activity using questionnaires. To determine whether this protocol is feasible, the investigators will examine participant recruitment and retention rates.

DETAILED DESCRIPTION:
Over the past two decades, society has encouraged people to be more physically active. As a result, most individuals are now aware of the positive effects of regular physical activity and have the intention to exercise. Yet, this intention is not sufficient, as exercise plans are often not executed. Despite gradually scaling up actions that promote physical activity over the years, people are actually becoming less active. From 2010 to 2016, the number of inactive adults has increased by 5% worldwide, currently affecting more than 1 in 4 adults (1.4 billion people). This gap between intention and action is a challenge that health professionals need to address in order to counteract the pandemic of physical inactivity.

Physical activity is one of the top contributors to health, reducing rates of cardiovascular disease, cancer, hypertension, diabetes, obesity, and depression. This wide spectrum of benefits is particularly important for older adults, who often suffer structural and functional deterioration across several physiological systems. Physical activity can reduce and delay the impact of this age-related deterioration in health and functional independence. However, in the Americas, more than 60% of older adults are physically inactive.

Current interventions to enhance physical activity in older adults rely mainly on reflective processes by providing rational information about the health benefits of a physically active lifestyle. From this perspective, changing conscious goals should lead to substantial behavioural change. Yet, meta-analyses indicate that these interventions are more effective in changing intentions than actual behaviour. Thus, new interventions targeting alternative processes are necessary to explore.

Recent work highlights that engagement in physical activity is governed not only by reflective processes, but also by automatic processes acting outside conscious awareness. For example, in active individuals, stimuli associated with physical activity attract attention, trigger positive affective reactions, and activate approach tendencies. These automatic reactions are thought to facilitate the translation of intention into action. From this perspective, physical inactivity is the result of an imbalance between strong negative automatic reactions to stimuli associated with physical activity and a relatively weaker intention to be physically active. This imbalance between reflective and automatic processes can be particularly pronounced in older adults, who are more likely to spontaneously associate physical activity with fear, pain, or discomfort felt during physical exercise. Therefore, older adults could be particularly responsive to and benefit the most from an intervention targeting the automatic reactions to physical activity and sedentary stimuli.

Interventions targeting automatic reactions to health-related stimuli have already proven to be successful in changing behaviour. For example, interventions have been used to retrain the automatic reaction to alcohol. Using a joystick, patients were repeatedly asked to avoid pictures on a screen that were related to alcohol and to approach pictures unrelated to alcohol. Results showed that adding to a regular treatment an intervention targeting cognitive bias reduced the relapse rates one year after treatment discharge by 9% to 13%. These interventions have also proven to be useful in impacting smoking, social anxiety, and eating behaviour.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Able to walk
* Able to communicate in English
* Able to travel to the University of Ottawa Lees Campus

Exclusion Criteria:

* Diagnosed neurological or psychiatric disorder
* Impaired motor function of the upper limbs
* Unable to understand task instructions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any and all self-identified genders are permitted to join this study.
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Determinants of Protocol Feasibility: Recruitment Rate and Retention Rate | From enrollment to the end of recruitment at 7 months
  The main purpose of this study is to determine whether the intervention protocol is feasible and thus the primary outcomes are recruitment rates, retention rates, and reasons for study dropout.

SECONDARY OUTCOMES:
Actigraph wGT3X-BT accelerometers for measuring daily step count | From enrollment to the end of recruitment at 7 months
  Participants will wear the a small research grade accelerometer on their right hip with support hardware supplied by the researchers to measure their daily step count. As a key measure of physical activity, this device will be worn for 1 week before intervention, after intervention, and once more 1 month after the intervention.
Approach Avoidance Task | From enrollment to the end of recruitment at 7 months
  The manikin approach avoidance task has been previously used to determine automatic attitudes towards physical activity and sedentary behaviour. It is a laptop-based task where participants move an avatar towards or away from an image of physical activity or sedentary behaviour. The task measures the reaction time that participants respond to each image type to determine whether they have biased tendencies towards a certain image.
6 Minute Walk Test | From enrollment to the end of recruitment at 7 months
  The 6 Minute Walk Test is a common measure to assess walking ability. The test is conducted by having the participant walk as far as possible on a 30m flat indoor course for a period of 6 minutes. Standardized encouragement will be provided at each minute. Total distance walked (meters) in 6 minutes will be documented. The major outcome is the distance walked during the 6 minutes.
Hand Dynamometer for Grip Strength | From enrollment to the end of recruitment at 7 months
  Grip strength will be assessed with the JAMAR Hand Dynamometer. Participants will perform the test using their reported dominant hand in a seated position with their elbow flexed 90 degrees. Two tests would be performed by each participant and the higher value (Kilogram*Force) will be recorded as hand grip strength.
World Health Organization Quality of Life Questionnaire (WHOQOL) | From enrollment to the end of recruitment at 7 months
  The scale assesses quality of life (QoL) over four domains: Physical Health (seven items), Psychological Health (six items), Social Relationships (three items), and Environmental Health (eight items). Scores for each item can range from one to five with higher scores indicating better QoL.
Affective and Instrumental Attitude Scale (ASIS) | From enrollment to the end of recruitment at 7 months
  This scale assesses participants' attitudes towards physical activity. It has four questions scored from one to seven assessing affective and instrumental attitudes. Scores nearer 1 indicate less affective/instrumental attitudes while scores nearer 7 indicate greater affective/instrumental attitudes.
Physical Effort Scale (PES) | From enrollment to the end of recruitment at 7 months
  This questionnaire asks about the participant's perceptions about physical effort, which is usually associated with increased heart rate and breathing. It consists of eight items ranging from one to five with higher scores indicating greater agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Kayne Park, PhD, Principal Investigator — University of Ottawa; Matthieu P Boisgontier, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Faculty of Health Sciences, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data from participants that were included in the final study report will be shared on an online repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD and supporting information will be available for an indefinite time on an online repository once the data collection is complete.
Access Criteria: All data of participants with full datasets collected in this study will be accessible after the data collection has completed.

REFERENCES:
- [Background] Veling, H., Becker, D., Liu, H., Quandt, J., & Holland, R. W. How go/no-go training changes behavior: A value-based decision-making perspective. Current Opinion in Behavioral Sciences. 2022;47:101206.
- [Background] Scott SH. Apparatus for measuring and perturbing shoulder and elbow joint positions and torques during reaching. J Neurosci Methods. 1999 Jul 15;89(2):119-27. doi: 10.1016/s0165-0270(99)00053-9. PMID 10491942
- [Background] Rhodes RE, McEwan, D, Rebar AL. Theories of physical activity behavior change: A history and synthesis of approaches. Psychology of Sport and Exercise. 2019;42:100-9.
- [Background] Marteau TM, Hollands GJ, Fletcher PC. Changing human behavior to prevent disease: the importance of targeting automatic processes. Science. 2012 Sep 21;337(6101):1492-5. doi: 10.1126/science.1226918. PMID 22997327
- [Background] Conroy DE, Hyde AL, Doerksen SE, Ribeiro NF. Implicit attitudes and explicit motivation prospectively predict physical activity. Ann Behav Med. 2010 May;39(2):112-8. doi: 10.1007/s12160-010-9161-0. PMID 20140542
- [Background] Chevance G, Bernard P, Chamberland PE, Rebar A. The association between implicit attitudes toward physical activity and physical activity behaviour: a systematic review and correlational meta-analysis. Health Psychol Rev. 2019 Sep;13(3):248-276. doi: 10.1080/17437199.2019.1618726. Epub 2019 Jun 12. PMID 31117901
- [Background] Cheval B, Tipura E, Burra N, Frossard J, Chanal J, Orsholits D, Radel R, Boisgontier MP. Avoiding sedentary behaviors requires more cortical resources than avoiding physical activity: An EEG study. Neuropsychologia. 2018 Oct;119:68-80. doi: 10.1016/j.neuropsychologia.2018.07.029. Epub 2018 Jul 26. PMID 30056055
- [Background] Cheval B, Sarrazin P, Isoard-Gautheur S, Radel R, Friese M. Reflective and impulsive processes explain (in)effectiveness of messages promoting physical activity: a randomized controlled trial. Health Psychol. 2015 Jan;34(1):10-9. doi: 10.1037/hea0000102. Epub 2014 Aug 18. PMID 25133840
- [Background] Cheval B, Boisgontier MP. The Theory of Effort Minimization in Physical Activity. Exerc Sport Sci Rev. 2021 Jul 1;49(3):168-178. doi: 10.1249/JES.0000000000000252. PMID 34112744
- [Background] Aulbach MB, Knittle K, Haukkala A. Implicit process interventions in eating behaviour: a meta-analysis examining mediators and moderators. Health Psychol Rev. 2019 Jun;13(2):179-208. doi: 10.1080/17437199.2019.1571933. Epub 2019 Feb 6. PMID 30676235